CLINICAL TRIAL: NCT03225157
Title: Observational Study of Hearing Loss and the Effects of Statin Drugs in Head and Neck Squamous Cell Carcinoma Patients Treated With Cisplatin Chemoradiation
Brief Title: Hearing Loss and the Effects of Statin Drugs in People With Head and Neck Squamous Cell Carcinoma Treated With Cisplatin Chemoradiation
Status: Completed | Type: Observational
Sponsor: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 170138; 17-DC-0138
Record Dates: First submitted 2017-07-20; First posted 2017-07-21 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Head and Neck Neoplasms; Hearing Disorder; Hyperlipidemia
Keywords: Audiogram; Statins; Drug Response; Cancer Treatment; Head and Neck Cancer; Natural History
MeSH Terms: conditions — Head and Neck Neoplasms; Hearing Disorders; Hyperlipidemias

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: adult patients with head and neck squamous cell carcinoma of the upper aerodigestive tract who will undergo cisplatin chemotherapy with concurrent radiation.

SUMMARY:
Background:

Cisplatin is a chemotherapy drug. It is used to treat head and neck squamous cell carcinoma (HNSCC) and other cancers. It can cause hearing loss for some people. It is not known how many people will get hearing loss from cisplatin. It is also not known what other factors might influence who gets hearing loss. Factors could include age, sex, noise exposure, and other drugs the person is taking. Statins are drugs used to lower cholesterol. Statins may also reduce cisplatin-induced hearing loss.

Objectives:

To see if statins reduce hearing loss in people getting cisplatin therapy to treat HNSCC. To find out how many people taking cisplatin get hearing loss from it. To find out if other factors might influence whether cisplatin causes hearing loss.

Eligibility:

People ages 18 and older who are getting treatment with cisplatin for HNSCC

Design:

Participants will be screened with a review of their medical records.

Participants will have 3 visits. These will be before the onset of cisplatin therapy, at about 4 weeks after they finish therapy, and about 6 months after they finish therapy. Each visit will include:

Medication history

Audiogram/hearing tests. Participants will wear headphones and indicate when they hear different sounds.

Questions about their noise exposure history and whether they have ringing in the ears

DETAILED DESCRIPTION:
Objectives:

* Primary: Determine whether head and neck cancer patients taking statin drugs for hyperlipidemia are at decreased risk of cisplatin-induced hearing loss.
* Secondary: Determine the incidence and severity of hearing loss in head and neck cancer patients undergoing low-dose, weekly cisplatin chemotherapy with concurrent radiation. Hearing loss with this more recent cisplatin regimen has not been thoroughly evaluated in the literature. Examine whether age, gender, pre-existing hearing loss, other medications, or comorbid medical conditions may be risk factors for cisplatin-induced hearing loss and/or the acquisition or progression of tinnitus in this patient population.

Study Population:

-Subjects will be adult patients with head and neck squamous cell carcinoma of the upper aerodigestive tract who will undergo cisplatin chemotherapy with concurrent radiation.

Design:

* Observational study
* 334 subjects will be enrolled.
* Subjects will complete a questionnaire to estimate the degree of prior noise exposure and impact on baseline hearing. Information on medical comorbidities, names and doses of current medications will be obtained from the medical record and verified at each subject visit.
* Subjects will complete self-administered audiograms using FDA-approved software from SHOEBOXTM Audiometry on a portable tablet (iPad) computer.
* Audiograms will be completed prior to commencing chemoradiation, within 4 weeks of completing treatment, and 6 months after completing treatment.
* Subjects will also complete a validated tinnitus questionnaire with each audiogram. A noise exposure history will be collected during the initial study visit and verified during subsequent visits. Any indicated changes to the subject s noise exposure history will be added to record.
* No investigational or experimental therapy will be given as part of this protocol.
* Audiograms will be performed at the Johns Hopkins Suburban Outpatient Center or the NIH Clinical Center.
* Two interim analyses will be conducted prior to study completion (after N=88 and N=176 subjects completing the protocol) to determine whether there are statistically significant differences in severity or incidence of hearing loss in subjects taking concurrent statin drugs vs. subjects who are not taking statin drugs.

Outcome Measures:

* Primary outcome measure: The primary outcome measure is the change in hearing sensitivity (as measured by the self-administered audiogram) between the pre-treatment (before cisplatin therapy) hearing test and the post-treatment (after completion of cisplatin therapy) audiogram. Hearing loss will be defined according to TUNE and ASHA criteria and will be compared in subjects taking statin drugs vs. subjects not taking statin drugs. Hearing status will be compared between audiograms collected at baseline (prior to treatment) to a repeated audiogram at the end of treatment (within 4 weeks of cisplatin protocol cessation).
* Secondary outcome measure: Secondary outcome measures include 1) changes in hearing sensitivity between the first post-cisplatin audiogram and the second post-cisplatin audiogram, and 2) changes in scores on the tinnitus questionnaire between the pre-treatment audiogram and the two post-treatment audiograms.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Adult patients over the age of 18.
* Patients with squamous cell carcinoma of the upper aerodigestive tract including the larynx, hypopharynx, oropharynx, and oral cavity who undergo treatment with concomitant cisplatin chemotherapy and intensity-modulated radiotherapy (IMRT) with curative intent.
* Patients treated with cisplatin chemoradiation either as primary/definitive or adjuvant (post-surgical) therapy.
* Subjects must be able and willing to self-administer their hearing test via the iPad following a brief tutorial with one-on-one instruction from a member of the study team or medical staff.
* Subjects must have hearing thresholds at or better than 80 dB SPL at 1, 2, and 4 kilohertz (kHz) at the time of their baseline audiogram.
* Subjects must have a Type A tympanogram.
* Subjects must be able to provide their own consent.

EXCLUSION CRITERIA:

* Patients with carcinoma of the nasopharynx or paranasal sinuses, who may have Eustachian tube dysfunction (with resultant conductive hearing loss) related to radiation treatment involving these anatomic subsites.
* Patients with active middle ear disease that is likely to influence the results of audiograms during the study, as determined by an Investigator who is an otolaryngologist. If a potential subject reports active middle ear disease, medical records will be reviewed by a study otolaryngologist to determine whether the patient should be excluded.
* Patients with cochlear implants will be excluded.
* Patients with a history of prior treatment with platinum chemotherapy drugs will be excluded.
* Patients who receive taxanes or other cytotoxic chemotherapy drugs in addition to cisplatin will be excluded. The standard of care is cisplatin as monotherapy for previously untreated HNSCC.
* Staff members of the NIDCD Sections that are headed by the PI and LAI will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be adult patients with head and neck squamous cell carcinoma of the upper aerodigestive tract who will undergo cisplatin chemotherapy with concurrent radiation.
Sampling Method: Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2017-11-03 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
Primary outcome measure: Determine whether head and neck cancer patients taking statin drugs for hyperlipidemia are at decreased risk of cisplatin-induced hearing loss. | 03/01/2022
  The primary outcome measure is the change in hearing sensitivity (as measured by the self-administered audiogram) between the pre-treatment (before cisplatin therapy) hearing test and the post-treatment (after completion of cisplatin therapy) audiogram. Hearing loss will be defined according to TUNE and ASHA criteria and will be compared in subjects taking statin drugs vs. subjects not taking statin drugs. Hearing status will be compared between audiograms collected at baseline (prior to treatment) to a repeated audiogram at the end of treatment (within 4 weeks of cisplatin protocol cessation).

SECONDARY OUTCOMES:
Determine the incidence and severity of hearing loss in head and neck cancer patients undergoing low-dose, weekly cisplatin chemotherapy with concurrent radiation. | 03/01/2022
  Secondary outcome measures include 1) changes in hearing sensitivity between the first post-cisplatin audiogram and the second post-cisplatin audiogram, and 2) changes in scores on the tinnitus questionnaire between the pre-treatment audiogram and the two post-treatment audiograms.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa L Cunningham, Ph.D., Principal Investigator — National Institute on Deafness and Other Communication Disorders (NIDCD)
Locations (2):
- United States (2):
  - Johns Hopkins Suburban Hospital, Bethesda, Maryland
  - National Institutes of Health Clinical Center, Bethesda, Maryland

REFERENCES:
- [Derived] Fernandez KA, Allen P, Campbell M, Page B, Townes T, Li CM, Cheng H, Garrett J, Mulquin M, Clements A, Mulford D, Ortiz C, Brewer C, Dubno JR, Newlands S, Schmitt NC, Cunningham LL. Atorvastatin is associated with reduced cisplatin-induced hearing loss. J Clin Invest. 2021 Jan 4;131(1):e142616. doi: 10.1172/JCI142616. PMID 33393488
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2017-DC-0138.html